CLINICAL TRIAL: NCT03161834
Title: LCCC 1642: Plasma Circulating Tumor DNA (ctDNA) Analyses in ER+ Metastatic Breast Cancer
Brief Title: Plasma Circulating Tumor DNA Analyses in ER+ Metastatic Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: IRB Study Closure
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1642; 16-2952 (Other: UNC IRB)
Record Dates: First submitted 2017-05-15; First posted 2017-05-22 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Breast Cancer
Keywords: DNA; Circulating tumor cells
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 mL blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational

SUMMARY:
The purpose of this study is to evaluate whether increased mutant ESR1 allele fraction in plasma ctDNA 3-6 weeks after initiating salvage endocrine therapy is predictive of progression free survival in patients with ER+ metastatic breast cancer.

DETAILED DESCRIPTION:
The primary objective of this 110 patient correlative biomarker study is to evaluate whether changes in mutant ESR1 allele fraction in plasma circulating tumor DNA (ctDNA) are predictive of progression-free survival in metastatic ER+ breast cancer patients who are receiving 2nd, 3rd, or 4th line systemic endocrine therapy. A secondary goal of this study is to explore the prevalence and kinetics of hotspot and non-hotspot ctDNA ESR1 mutations in this patient population, prior to initiating a new line of endocrine therapy as well as upon clinical progression, to identify potential mechanisms of resistance. Although initially to be opened at UNC Chapel Hill, our goal is to expand enrollment to include Rex Cancer Center in Raleigh, North Carolina, and collaborating institutions through the Translational Breast Cancer Research Consortium.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Female gender
* Biopsy proven diagnosis of breast cancer
* Stage IV disease diagnosed either by radiographic studies or biopsy
* ER+ by immunohistochemistry on primary and/or metastatic tissue biopsy (>10%)
* HER2 non-amplified (1+ or below by immunohistochemistry, and/or Her2 FISH <2 HER2-to-CEP17 ratio)
* Progressed on at least one prior line of endocrine therapy for metastatic disease
* Three or fewer prior endocrine-containing therapies for recurrent/metastatic disease
* Two or fewer prior lines of cytotoxic chemotherapy for recurrent/metastatic disease
* Plans to initiate 2nd, 3rd, or 4th line endocrine therapy for metastatic disease
* Recent re-staging scans within 4 weeks of study enrollment, with radiographically identifiable disease
* No concurrent or prior diagnosis of malignancy other than breast cancer for the past 5 years. Patients with a history of in situ cancer or basal or localized squamous cell skin cancer remain eligible
* Intends to pursue treatment as well as clinical and radiographic follow-up at UNC Health Care
* Signed an institutional review board (IRB)-approved informed consent document for this protocol and HIPAA consent form

Exclusion Criteria:

* < 18 years of age
* Tissue biopsies that support the presence of both ER+ and ER- metastatic breast cancer in the same patient
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Pregnant or lactating women

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with metastatic breast cancer
Study Population: Females with ER+ metastatic breast cancer receiving 2nd, 3rd, or 4th line systemic endocrine therapy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival Prediction | Through study completion, an average of 3-6 weeks
  To evaluate whether increased mutant ESR1 allele fraction in plasma ctDNA 3-6 weeks after initiating salvage endocrine therapy is predictive of progression free survival in patients with ER+ metastatic breast cancer.

SECONDARY OUTCOMES:
DNA Analysis of Hotspot Mutation Prevalence | Through study completion, an average of 3-6 weeks
  To evaluate the overall spectrum and prevalence of hotspot and non-hotspot ESR1 mutations in plasma ctDNA prior to initiating 2nd, 3rd, or 4th endocrine therapy and after clinical disease progression.
DNA Analysis of Mutation and Radiographic Response Correlation | Through study completion, an average of 3-6 weeks
  Exploratory analysis of whether changes in mutant ESR1 allele fraction in plasma ctDNA at the time of re-staging scans correlates with radiographic response.

CONTACTS AND LOCATIONS:
Overall Officials: Gaorav P Gupta, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill Cancer Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials